CLINICAL TRIAL: NCT02801656
Title: Fecal Microbiota Transplantation for Primary Therapy in Clostridium Difficile Diarrhea - A Placebo-blinded Randomized Clinical Trial
Brief Title: Fecal Microbiota Transplantation for Primary Clostridium Difficile Diarrhea
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Not funded
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Peter Daley, Assistant Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MUN-02
Record Dates: First submitted 2016-06-09; First posted 2016-06-16 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Clostridium Difficile
MeSH Terms: interventions — Fecal Microbiota Transplantation; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal Microbiota Transplantation (Experimental): Oral, encapsulated fecal microbiota transplantation
  Interventions: Biological: Fecal Microbiota Transplantation; Drug: Vancomycin Placebo
- Vancomycin (Active Comparator): 125 mg po qid x 10 days
  Interventions: Drug: Vancomycin; Biological: Fecal Microbiota Transplantation Placebo

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — Oral, encapsulated FMT
  Other Names: Stool Transplant
  Arms: Fecal Microbiota Transplantation
Drug: Vancomycin — Vancomycin po 125 mg qid x 10 days
  Other Names: Vancocin
  Arms: Vancomycin
Biological: Fecal Microbiota Transplantation Placebo — Matching placebo to FMT
  Other Names: Stool Transplant Placebo
  Arms: Vancomycin
Drug: Vancomycin Placebo — Matching placebo to Vancomycin
  Other Names: Vancocin Placebo
  Arms: Fecal Microbiota Transplantation

SUMMARY:
Clostridium difficile associated diarrhea (CDAD) is a significant cause of morbidity and mortality, caused by loss of healthy gut flora. Conventional treatment uses antibiotics to kill Clostridium difficile. A novel treatment uses replacement of gut flora by fecal microbiota transplant (FMT). Randomized trials have established safety and efficacy of FMT in recurrent CDAD, but no trial has used FMT for primary CDAD. This study will randomize patients to oral encapsulated FMT or oral Vancomycin.

DETAILED DESCRIPTION:
Patients with primary CDAD will be approached for consent and randomized equally to two arms: oral FMT with oral Vancomycin placebo, or oral FMT placebo with oral Vancomycin. FMT will be prepared from anonymous donors screened according to Health Canada guidelines and stored frozen.

ELIGIBILITY:
Inclusion Criteria:

* life expectancy > 3 months, 3 or more unformed stools in 24 hours prior to randomization, positive stool test within 72 hours of randomization

Exclusion Criteria:

* pregnancy, previous stool test positive within 12 months, toxic megacolon or ileus, already received >4 doses of treatment for current episode, inflammatory bowel disease, gastrointestinal surgery within 90 days of randomization (except appendectomy or cholecystectomy), documented aspiration of gastric contents within 90 days of randomization, requirement for treatment with oral probiotics, opiates, loperamide or diphenoxylate during the study duration, anticipated use of antibiotics for any reason during the study duration, known non-CDAD concurrent gastrointestinal infection, concurrent enrollment in another clinical trial for any reason, intolerance or hypersensitivity to Vancomycin, anaphylactic reaction to any food, current induction chemotherapy, HIV infection with Cluster of Differentiation 4 (CD4) count <200, or any medical or non-medical condition considered by the investigator to preclude participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Cure of diarrhea without recurrence in intention to treat population | 56 days
  Cure is defined as less than 3 bowel motions per day for 2 consecutive days during the 10 day treatment period. Recurrence is defined as 3 or more bowel motions within one day during the follow-up period.
Adverse Events | 56 days
  Number of participants with treatment-related adverse events as defined by the Medical Dictionary for Regulatory Activities.

SECONDARY OUTCOMES:
Efficacy: Cure of diarrhea without recurrence in a per protocol population | 56 days
  Cure is defined as less than 3 bowel motions per day for 2 consecutive days during the 10 day treatment period. Recurrence is defined as 3 or more bowel motions within one day during the follow-up period.
Efficacy: cure of diarrhea in intention to treat and per protocol populations | 10 days
  Cure is defined as less than 3 bowel motions per day for 2 consecutive days during the 10 day treatment period.
Efficacy: time to cure of diarrhea | 56 days
  Cure is defined as less than 3 bowel motions per day for 2 consecutive days during the 10 day treatment period.
Efficacy: Health status questionnaire | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Daley, MD FRCPC, Principal Investigator — Memorial University
Locations (1):
- Health Sciences Centre, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: Yes
After analysis is completed, data will be released